CLINICAL TRIAL: NCT04833972
Title: Eliciting Perceived Norms About Substance Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Alexander Tsai, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2013P000395_3
Record Dates: First submitted 2021-04-01; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Tobacco Use; Alcohol Drinking
MeSH Terms: conditions — Tobacco Use; Alcohol Drinking | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Study participants are randomly assigned to be read survey questions with slight changes in the wording of the response options. Neither study participants nor outcomes assessors are provided with information about "treatment" assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: V1: Binary Response Options (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. Each question in this version of the survey questionnaire has binary (yes/no) response options.
  Interventions: Other: Survey questionnaire
- Experimental: V2: Categorical Response Options (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. Each question in this version of the survey questionnaire has categorical response options: all or almost all; more than half, but fewer than 90%; fewer than half, but more than 10%; very few, or no one
  Interventions: Other: Survey questionnaire
- Experimental: V3: Open-Ended Numerical Estimate (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. Each question in this version of the survey questionnaire permits the study participant to provide an open-ended numerical estimate.
  Interventions: Other: Survey questionnaire

INTERVENTIONS:
Other: Survey questionnaire — Each version of the questionnaire has the same questions about perceived norms about substance use in the community but differs in how the response options are offered.

SUMMARY:
Survey experiment to elicit perceived norms about substance use

DETAILED DESCRIPTION:
Health behaviors and health risk behaviors are known to be associated with the extent to which one perceives these behaviors as normative. The canonical example of this phenomenon is taken from the U.S. literature, which has robustly shown that undergraduate students on college campuses tend to drink more heavily and frequently if they believe their classmates drink heavily and frequently, irrespective of their classmates' actual levels and frequency of use. However, there remains little systematic understanding about the best ways to elicit these perceived norms through survey-based research studies. This randomized survey experiment compares different ways of eliciting perceived norms.

ELIGIBILITY:
Inclusion Criteria:

* All adults who consider Nyakabare their primary place of residence and who are capable of providing consent

Exclusion Criteria:

* Minors younger than 18 years of age, with the exception of emancipated minors
* Persons who do not consider Nyakabare Parish their primary place of residence, e.g., persons who happen to be visiting Nyakabare at the time of the survey or who own a home in Nyakabare but spend most of their time outside the parish
* Persons with psychosis, neurological damage, acute intoxication, or other cognitive impairment (all of which are determined informally in the field by non-clinical research staff in consultation with a supervisor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1553 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Perception of Tobacco Use Frequency Among Men | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most men in your cell in this parish smoked cigarettes four or more times per week in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Tobacco Use Frequency Among Women | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most women in your cell in this parish smoked cigarettes four or more times per week in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Use Frequency Among Men | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most men in your cell in this parish taken alcohol four or more times per week in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Use Frequency Among Women | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most women in your cell in this parish taken alcohol four or more times per week in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol-Related Blackouts Among Men | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 30 days)
  "According to your perception, have most men in your cell in this parish been unable to remember what happened the night before at least once as a result of them taking alcohol in the past 30 days?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol-Related Blackouts Among Women | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 30 days)
  "According to your perception, have most women in your cell in this parish been unable to remember what happened the night before at least once as a result of them taking alcohol in the past 30 days?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol-Related Spousal Problems Among Men | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 30 days)
  "According to your perception, have most men in your cell in this parish quarreled after taking alcohol with their spouse or main partner if they have one in the past 30 days?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol-Related Spousal Problems Among Women | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 30 days)
  "According to your perception, have most women in your cell in this parish quarreled after taking alcohol with their spouse or main partner if they have one in the past 30 days?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Intoxication Among Men | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 30 days)
  "According to your perception, have most men in your cell in this parish experienced drunkenness or intoxication on 3 or more days in the past 30 days?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Intoxication Among Women | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 30 days)
  "According to your perception, have most women in your cell in this parish experienced drunkenness or intoxication on 3 or more days in the past 30 days?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Use Financial Harms Among Men | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most men in your cell in this parish had a harmful effect on their household's finances due to them taking alcohol in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Use Financial Harms Among Women | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most women in your cell in this parish had a harmful effect on their household's finances due to them taking alcohol in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Spending Among Men | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most men in your cell in this parish spent more than 35,000 USh on any kind of alcohol in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Spending Among Women | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most women in your cell in this parish spent more than 35,000 USh on any kind of alcohol in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Binge Use Frequency Among Men | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most men in your cell in this parish taken 6 or more drinks in a single morning, afternoon, or night in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)
Perception of Alcohol Binge Use Frequency Among Women | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate, and participants are asked about the past 12 months)
  "According to your perception, have most women in your cell in this parish taken 6 or more drinks in a single morning, afternoon, or night in the past 12 months?" (single item, culturally adapted and developed for this study; categorical response options)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No